CLINICAL TRIAL: NCT02571400
Title: Prevalence and Predictors of Prolonged Post-surgical Opioid Use: a Prospective Observational Cohort Study
Status: Completed | Type: Observational
Sponsor: University of Notre Dame Australia (Other)
Collaborators: St Vincent's Hospital, Sydney (Other)
Responsible Party: Principal Investigator, Natasha Stark, Medical student, University of Notre Dame Australia
Other Study IDs: UNDAustralia
Record Dates: First submitted 2015-10-05; First posted 2015-10-08 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Opioid Use Disorders; Opioid-related Disorders; Surgery; Pain, Postoperative; Post-operative Complications; Opiate Addiction
Keywords: Risk; Opioid analgesics; Opioid-related disorders; Surgery; Post-operative care; Post-operative period; Post-operative complications; Opioid Use disorders; Pain, post-operative; Opiate Addiction
MeSH Terms: conditions — Opioid-Related Disorders; Pain, Postoperative | interventions — Postoperative Period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients scheduled to undergo surgery: Patients scheduled to undergo surgery at St Vincent's Private Hospital Sydney
  Interventions: Other: Continued use of opioid analgesics >90 days post-surgery

INTERVENTIONS:
Other: Continued use of opioid analgesics >90 days post-surgery — Exposure of interest: continued use of opioid analgesics >90 days post-surgery

SUMMARY:
Post-surgical opioid prescribing intended for the short-term management of acute pain may lead to long-term opioid use, and its associated harms. This study was undertaken to determine the prevalence of prolonged post-surgical opioid use, and patient-related factors associated with prolonged post-surgical opioid use.

DETAILED DESCRIPTION:
There are growing concerns that surgery is a risk factor for chronic opioid use. Existing studies suggest that post-surgical opioid prescribing intended for the short-term management of acute pain may result in unintended long-term opioid use for a small, but meaningful number of patients.

Increasing numbers of patients are discharged from hospital post-surgery with opioids for the management of their acute post-surgical pain. Opioids have proven efficacy for the management of acute post-surgical pain, but can cause significant harm when used long-term for non-cancer pain. Evidence suggests that post-surgical opioid use continues in some patients for years after surgery.

Identification of patients at risk of prolonged opioid use after surgery may assist in reducing the adverse outcomes associated with long-term opioid use. Pre-operative risk stratification tools may be of use in identifying surgical patients at risk of long-term opioid use. Validated tools are widely used to identify patients at high risk of opioid misuse in the chronic pain setting, but currently there is no optimal method to predict patients at risk of chronic opioid use after surgery.

Existing studies have found that a wide range of patient characteristics and psychiatric comorbidities are associated with long-term opioid use in a post-surgical setting.

There are 5 primary study procedures in the investigators research project:

1. Enrolment in the study: Subjects will be recruited and enrolled at the pre-operative admission clinic and day surgery unit at St Vincent's Private Hospital, Sydney. This study aims to enrol 1000 patients.
2. Informed consent: Patients who meet inclusion criteria, and agree to enrol in the study will be asked to read and sign an informed consent document.
3. Initial questionnaire: Trained nursing staff will administer an initial questionnaire to all patients participating in the study. This questionnaire will gather data regarding potential predictors of delayed opiate cessation including age, sex, operation type, pre-operative opioid use, depression traits, anxiety traits, addictive traits, perceived susceptibility to addiction, average hours of sleep per night, history of chronic pain, and perceived general health.
4. Follow-up questionnaire: At approximately 90 days post-surgery, a follow-up questionnaire will be administered to all enrolled subjects via phone call or email. This questionnaire will determine current pain scores and details regarding current pain medication usage.
5. Statistical analysis: Once data collection is complete, identifying details will be removed, and data will be entered into a password-protected electronic database. The investigators will analyse data from all patients and determine the prevalence of delayed opioid cessation, and which questionnaire items independently predict delayed opioid cessation.

The investigators primary study objective is to determine the prevalence of prolonged post-surgical opioid use, defined by our study as patients taking opioids >90 days post-surgery. The investigators secondary objective is to identify patient-related factors that are independently associated with prolonged post-surgical opioid use. These factors may be used to develop a pre-operative screening tool for patients undergoing surgery, in order to assign a level of risk for chronic post-surgical opioid use.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Able to give written informed consent
* Willing to participate and comply with the study
* Scheduled to undergo surgery at St Vincent's Private Hospital, and attending the pre-admission clinic or day surgery unit

Exclusion Criteria:

* Opioid tolerant patients (patients who are chronically receiving opioid analgesics on a daily basis)
* Scheduled to undergo surgery relating to malignancy
* Surgical procedures completed under local anaesthetic
* Minimally invasive procedures including gastroscopy, colonoscopy, bronchoscopy, cardioversion or transoesophageal echo
* Patients who were unable to complete study questionnaires due to psychological illness, medical condition or significant language barrier were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pre-Admission Clinic, St Vincent's Private Hospital (pre-operative assessment unit) Day Surgery Unit, St Vincent's Private Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1013 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Continued opioid use | 90 days post-surgery
  Subjects will be recruited to the study from October 2015 to March 2016, prior to their elective surgical procedure. All subjects will be contacted by investigators at 90 days post-surgery. At this point, they will be asked questions regarding their current analgesic use. This will enable us to calculate the prevalence of continued opioid use at ≥90 days post-surgery. Data collection will be complete by June 2016.

SECONDARY OUTCOMES:
Pain scores (score/10) | 90 days post-surgery
  Subjects will be recruited to the study from October 2015 to March 2016, prior to their elective surgical procedure. All subjects will be contacted by investigators at 90 days post-surgery. At this point, they will be asked questions regarding their current pain scores out of 10. Data collection will be complete by June 2016.
Presence of pre-operative potential predictors of delayed opioid cessation | 90 days post-surgery
  Subjects will be recruited to the study from October 2015 to March 2016, prior to their elective surgical procedure. Subjects will complete a single questionnaire prior to surgery which will collect data including their age, sex, operation type, pre-operative opioid use, depression traits, anxiety traits, addictive traits, perceived susceptibility to addiction, average hours of sleep per night, history of chronic pain, and perceived general health.
  The investigators will compare subjects with and without delayed opioid cessation to see which questionnaire items were able to independently predict continued opioid use >90 days post-surgery. Data collection will be complete by June 2016.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Stevens, MBChB, Principal Investigator — St Vincent's Hospital, Sydney
Locations (1):
- St Vincent's Private Hospital, Sydney, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hollingworth SA, Gray PD, Hall WD, Najman JM. Opioid analgesic prescribing in Australia: a focus on gender and age. Pharmacoepidemiol Drug Saf. 2015 Jun;24(6):628-36. doi: 10.1002/pds.3767. Epub 2015 Apr 1. PMID 25845470
- [Background] Chou R, Fanciullo GJ, Fine PG, Adler JA, Ballantyne JC, Davies P, Donovan MI, Fishbain DA, Foley KM, Fudin J, Gilson AM, Kelter A, Mauskop A, O'Connor PG, Passik SD, Pasternak GW, Portenoy RK, Rich BA, Roberts RG, Todd KH, Miaskowski C; American Pain Society-American Academy of Pain Medicine Opioids Guidelines Panel. Clinical guidelines for the use of chronic opioid therapy in chronic noncancer pain. J Pain. 2009 Feb;10(2):113-30. doi: 10.1016/j.jpain.2008.10.008. PMID 19187889
- [Background] Hah JM, Mackey S, Barelka PL, Wang CK, Wang BM, Gillespie MJ, McCue R, Younger JW, Trafton J, Humphreys K, Goodman SB, Dirbas FM, Schmidt PC, Carroll IR. Self-loathing aspects of depression reduce postoperative opioid cessation rate. Pain Med. 2014 Jun;15(6):954-64. doi: 10.1111/pme.12439. PMID 24964916
- [Background] Singh JA, Lewallen DG. Predictors of use of pain medications for persistent knee pain after primary Total Knee Arthroplasty: a cohort study using an institutional joint registry. Arthritis Res Ther. 2012 Nov 16;14(6):R248. doi: 10.1186/ar4091. PMID 23157942
- [Background] Singh JA, Lewallen DG. Predictors of pain medication use for arthroplasty pain after revision total knee arthroplasty. Rheumatology (Oxford). 2014 Oct;53(10):1752-8. doi: 10.1093/rheumatology/ket443. Epub 2014 Jan 22. PMID 24459220
- [Background] Carroll I, Barelka P, Wang CK, Wang BM, Gillespie MJ, McCue R, Younger JW, Trafton J, Humphreys K, Goodman SB, Dirbas F, Whyte RI, Donington JS, Cannon WB, Mackey SC. A pilot cohort study of the determinants of longitudinal opioid use after surgery. Anesth Analg. 2012 Sep;115(3):694-702. doi: 10.1213/ANE.0b013e31825c049f. Epub 2012 Jun 22. PMID 22729963
- [Background] Singh JA, Lewallen D. Predictors of pain and use of pain medications following primary Total Hip Arthroplasty (THA): 5,707 THAs at 2-years and 3,289 THAs at 5-years. BMC Musculoskelet Disord. 2010 May 13;11:90. doi: 10.1186/1471-2474-11-90. PMID 20462458
- [Background] Sun EC, Darnall BD, Baker LC, Mackey S. Incidence of and Risk Factors for Chronic Opioid Use Among Opioid-Naive Patients in the Postoperative Period. JAMA Intern Med. 2016 Sep 1;176(9):1286-93. doi: 10.1001/jamainternmed.2016.3298. PMID 27400458
- [Background] Macintyre PE, Huxtable CA, Flint SL, Dobbin MD. Costs and consequences: a review of discharge opioid prescribing for ongoing management of acute pain. Anaesth Intensive Care. 2014 Sep;42(5):558-74. doi: 10.1177/0310057X1404200504. PMID 25233168
- [Background] Alam A, Gomes T, Zheng H, Mamdani MM, Juurlink DN, Bell CM. Long-term analgesic use after low-risk surgery: a retrospective cohort study. Arch Intern Med. 2012 Mar 12;172(5):425-30. doi: 10.1001/archinternmed.2011.1827. PMID 22412106
- [Background] Clarke H, Soneji N, Ko DT, Yun L, Wijeysundera DN. Rates and risk factors for prolonged opioid use after major surgery: population based cohort study. BMJ. 2014 Feb 11;348:g1251. doi: 10.1136/bmj.g1251. PMID 24519537
- [Background] Goesling J, Moser SE, Zaidi B, Hassett AL, Hilliard P, Hallstrom B, Clauw DJ, Brummett CM. Trends and predictors of opioid use after total knee and total hip arthroplasty. Pain. 2016 Jun;157(6):1259-1265. doi: 10.1097/j.pain.0000000000000516. PMID 26871536
- [Background] Quinn PD, Hur K, Chang Z, Krebs EE, Bair MJ, Scott EL, Rickert ME, Gibbons RD, Kroenke K, D'Onofrio BM. Incident and long-term opioid therapy among patients with psychiatric conditions and medications: a national study of commercial health care claims. Pain. 2017 Jan;158(1):140-148. doi: 10.1097/j.pain.0000000000000730. PMID 27984526